CLINICAL TRIAL: NCT04379648
Title: Assessment of Dissociative Traumatic Disorders
Acronym: TEDI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Januel (Other)
Responsible Party: Sponsor-Investigator, Januel, Clinical research unit manager, Centre hospitalier de Ville-Evrard, France
Organization: Centre hospitalier de Ville-Evrard, France (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 10477M-TEDI
Record Dates: First submitted 2020-04-29; First posted 2020-05-07 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Diagnostic Self Evaluation

STUDY DESIGN:
Intervention Model Description: All patients with a diagnosis of Post Traumatic Stress Disorder will be seen by a physician psychiatrist or psychologist who will introduce them to the study. They will be given an information letter and a consent form. If patients agree to participate in the study, and after signing the consent form, they will be included and will complete the assessment scales.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Posttraumatic stress disorder (Other): cohort of patients with Posttraumatic stress disorder PTSD
  Interventions: Other: self-assessment and hetero-assessment

INTERVENTIONS:
Other: self-assessment and hetero-assessment — Self assessment for the passing of the following rating scales CTQ-SF36-ITQ-PCL5-DES Hetero-assessment for the pasing of the following rating scales DDIS FR and medical interview

SUMMARY:
More than 70% of ambulatory patients with IDD have attempted suicide (APA, 2015). This disorder, as well as all the disorders on the dissociation spectrum, must therefore be clarified and better diagnosed.

The goal of this research is :

1. to assess the prevalence of dissociative disorders using specific tools in patients suffering from PTSD.
2. to validate the French version of the DDIS interview (Ross, 1997) that the investigators have translated.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with PTSD according to DSM 5 criteria
* Over 18 years of age
* Informed consent signed

Exclusion Criteria:

* Neurological disorders
* Serious and/or unstable somatic pathologies
* Patient not affiliated with social security
* Patient hospitalized under restraint in psychiatric care by decision of the state representative or in psychiatric care at the request of a third party
* Patient under guardianship
* Patient participating in parallel in another biomedical research
* Change of antidepressant in the last three months
* Patient not mastering the French language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-02-05 (Actual); Primary Completion 2020-09-05 (Estimated); Study Completion 2021-09-05 (Estimated)

PRIMARY OUTCOMES:
Post Traumatic Stress | 1 year
  assessment of the prevalence of dissociative disorders in a cohort of patients with PTSD

CONTACTS AND LOCATIONS:
Overall Officials: Khalid KALALOU, Psychiatrist, Principal Investigator — EPS Ville Evrard
Locations (1):
- Youcef BENCHERIF, Neuilly-sur-Marne, Île-de-France Region, France